CLINICAL TRIAL: NCT05195177
Title: Nerve Excitability Testing Protocol to Efficiently Induce Itch
Brief Title: Testing Protocol to Efficiently Induce Itch
Acronym: ELIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Jenny Tigerholm, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-2020001 4-sub-project
Record Dates: First submitted 2021-11-23; First posted 2022-01-18 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Drug: Anti-histamine cream 1 hour; Drug: Local anesthetic cream 1 hour

INTERVENTIONS:
Drug: Anti-histamine cream 1 hour — At the start of session 1, one area of the middle forearms of the participant will be located (4x4cm). On the area, anti-histamine cream will be applied for approximately 1 hour.
Drug: Local anesthetic cream 1 hour — At the start of session 2, one area of the middle forearms of the participant will be located (4x4cm). On the area, local anesthetic cream (2.5% lidocain/2.5 prilocaine) will be applied for approximately 1 hour.

SUMMARY:
This subproject aims to evaluate a new nerve excitability protocol to induce itch in healthy controls by electrical stimulation. Itch has many similarities with pain, and the nerve fibers that mediate the two sensations probably have the same morphological and excitability properties. The method used in this project will be the same as our research group uses for studying nociceptor fibers (PTT technique), but the focus is on the itch sensation. Since the itch fibers also terminate in the epidermis, our PTT technique should also be able to activate itch fibers, similar to pain fibers. If itch could be effectively induced by electrical stimulation, this would generate a valuable tool for studying itch in healthy controls. The sub-project takes place in 2 sessions (2 hours each).

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women in the age 18-80 years who speak and understand

Exclusion Criteria:

* Pregnancy or breast feeding
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous and present neurologic, musculoskeletal or mental illnesses (e.g., epilepsy, neuropathy, fibromyalgia and depression)
* Skin diseases
* Past history of conditions possibly leading to neuropathy
* Inability to cooperate
* Current use of medications that may affect the study, e.g., analgesics
* Previous traumatic experience of an electrical accident
* Consumption of alcohol or painkillers within the last 24 hours
* Participation in other pain studies throughout the study period
* Patients with cardiac diseases (e.g., pacemaker).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Perception threshold for pulse shape 1 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 1. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 2 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 2. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 3 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 3. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 4 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 4. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 1 when antihistamine cream has been applied | This outcome measurement will be estimated during session one. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 1 when anti-histamine cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 2 when anti-histamine cream has been applied | This outcome measurement will be estimated during session one. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 2 when anti-histamine cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 3 when anti-histamine cream has been applied | This outcome measurement will be estimated during session one. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 3 when anti-histamine cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 4 when anti-histamine cream has been applied | This outcome measurement will be estimated during session one. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 4 when anti-histamine cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 1 when local anaesthetic cream has been applied | This outcome measurement will be estimated during session two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 1 when local anaesthetic cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 2 when local anaesthetic cream has been applied | This outcome measurement will be estimated during session two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 2 when local anaesthetic cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 3 when local anaesthetic cream has been applied | This outcome measurement will be estimated during session two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 3 when local anaesthetic cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Perception threshold for pulse shape 4 when local anaesthetic cream has been applied | This outcome measurement will be estimated during session two. The outcome measure takes approximately 5 minutes to estimate.
  The perception threshold will be estimated for the electrical stimuli with pulse shape 4 when local anaesthetic cream has been applied for approximately an hour. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.
Sensation for pulse 1 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The investigator will ask the participant to rate the sensation of electrical stimulation with pulse 1 for the three different conditions. The conditions are: control (not active cream), antihistamine cream, and local anesthetic cream. The scale is 0-10 for the three sensations touch, itch, and pain. Zero means no sensation, and ten is the worst pain/touch/itch imaginable.
Sensation for pulse 2 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The investigator will ask the participant to rate the sensation of electrical stimulation with pulse 2 for the three different conditions. The conditions are: control (not active cream), antihistamine cream, and local anesthetic cream. The scale is 0-10 for the three sensations touch, itch, and pain. Zero means no sensation, and ten is the worst pain/touch/itch imaginable.
Sensation for pulse 3 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The investigator will ask the participant to rate the sensation of electrical stimulation with pulse 3 for the three different conditions. The conditions are: control (not active cream), antihistamine cream, and local anesthetic cream. The scale is 0-10 for the three sensations touch, itch, and pain. Zero means no sensation, and ten is the worst pain/touch/itch imaginable.
Sensation for pulse 4 | This outcome measurement will be estimated during sessions one and two. The outcome measure takes approximately 5 minutes to estimate.
  The investigator will ask the participant to rate the sensation of electrical stimulation with pulse 4 for the three different conditions. The conditions are: control (not active cream), antihistamine cream, and local anesthetic cream. The scale is 0-10 for the three sensations touch, itch, and pain. Zero means no sensation, and ten is the worst pain/touch/itch imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tigerholm, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Aalborg Ø, Denmark